CLINICAL TRIAL: NCT00398333
Title: Randomized Controlled, Open-label, Pilot Study to Assess the Effectiveness of a Nutritional Supplementation Enriched With Eicosapentaenoic Acid on Chemotherapy Tolerance in Patients With Advanced Colorectal Cancer
Brief Title: Study to Assess the Effectiveness of a Omega-3 Enriched Supplement on Chemotherapy Tolerance in Colon Cancer Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Impossibility to accomplish the sample size in assigned time.
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Pere Leyes, Specialist, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EPA-05; EPA-05/ ACA-SPAI-05-05 (Other: Hospital Clinic de Barcelona's Ethics Committee)
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Neoplasms; Eicosapentaenoic Acid; Quality of Life; Nutritional Status
MeSH Terms: conditions — Colorectal Neoplasms

ARMS (2):
- Eicosapentaenoic acid enriched nutritional supplement (Experimental)
  Interventions: Dietary Supplement: Eicosapentaenoic acid enriched nutritional supplement
- No supplementation (No Intervention)

INTERVENTIONS:
Dietary Supplement: Eicosapentaenoic acid enriched nutritional supplement — Oral intake of nutritional supplementation: a maximum of 480 mL or a minimum of 240 mL daily during the first 3 months of the study.
  Other Names: Prosure
  Arms: Eicosapentaenoic acid enriched nutritional supplement

SUMMARY:
The purpose of this study is to determine if a nutritional supplement enriched in omega-3 fatty acids is effective in improving the tolerance to chemotherapy treatment and improves quality of life.

DETAILED DESCRIPTION:
Colorectal cancer is one of the main causes of mortality in western countries. It is considered that in case of colorectal carcinoma, the frequency of weight loss at the moment of diagnosis is 54%. Undernourishment affects negatively the course of the illness and it confers a worse prognostic, increasing the morbidity and the mortality, while it entails an impairment in the quality of life of the patient.

There is a narrow relationship in the oncologic pathology between undernourishment and the pathology itself, drawing a common syndrome called cancerous cachexia. It is usual that patients subjected to chemotherapy present nutritional alterations due to the treatments' side effects.

With this study we want to assess the efficacy of a nutritional intervention with supplementation enriched in EPA to improve the tolerance to the antineoplastic treatment. As an index of tolerability to the chemotherapy treatment, it will be used the variation of changes in quality of life evaluated through the questionnaire EORTC QLQ-C30, using the parameters of global quality of life and physical function.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed of metastatic colon adenocarcinoma that are going to receive first line chemotherapy treatment in the oncology day hospital.
* Age over 18 years old.

Exclusion Criteria:

* Patients diagnosed of colon cancer are receiving second line chemotherapy.
* Antecedents of other malignant tumors with the exception of basocellular epithelioma.
* Chronic renal failure (Creatinine > 1.7).
* Previous diabetes mellitus.
* Obesity (IMC > 30)
* Medical conditions that imply hepatic encephalopathy, or ascites.
* Severe malnutrition according to the classification of the Subjective Global Assessment (SGA) or a BMI < 16.5.
* Major psychiatric disorder.
* Patients receiving enteral or parenteral nutrition.
* Contraindications for the indication of the nutritional supplement: Galactosemia.
* Seafood or seafood byproducts allergy.
* Patients taking drugs that affect the metabolism (anabolic steroids, orexigenic agents...).
* Absence of the informed consent form signed by the patient.
* Any patient who has disability to comply with the treatment or who has inability according to the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of a nutritional intervention with supplementation enriched in EPA to improve the tolerance to the antineoplastic treatment, using the variation in quality of life changes as the tolerability index. | 3 months

SECONDARY OUTCOMES:
To assess the influence of the nutritional status over the tolerance to the antineoplastic treatment. | 6 months
To assess the effect of a nutritional supplement over the nutritional status of the patient with disseminated neoplastic illness. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pere Leyes, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Catalonia, Spain

REFERENCES:
- [Result] Trabal J, Leyes P, Forga M, Maurel J. Potential usefulness of an EPA-enriched nutritional supplement on chemotherapy tolerability in cancer patients without overt malnutrition. Nutr Hosp. 2010 Sep-Oct;25(5):736-40. PMID 21336429